CLINICAL TRIAL: NCT06307847
Title: A Multi-center, Randomized, Double-Blinded, Active Controlled, Non-Inferiority, Phase III Clinical Trial to Evaluate Efficacy and Safety of SP5M001 Inj. as Compared to Synovian Inj. in Patients With Mild to Moderate Knee Osteoarthritis
Brief Title: Pivotal Study to Evaluate Efficacy and Safety of SP5M001 Inj. as Compared to Synovian Inj. in Patients With Mild to Moderate Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-HA-003
Record Dates: First submitted 2024-02-13; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis Thumb
Keywords: osteoarthritis, Knee; Intra-articular injection; hexamethylenediamine; Cross-linked hyaluronate
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP5M001 inj (Experimental): SP5M001 inj 5 ml pre-filled syringe into Knee joint cavity of osteoarthritis patients
  Interventions: Drug: SP5M001 inj
- Synovian inj (Active Comparator): Synovian inj 3 ml pre-filled syringe into Knee joint cavity of osteoarthritis patients
  Interventions: Drug: Synovian inj

INTERVENTIONS:
Drug: SP5M001 inj — pre-filled syringe
  Arms: SP5M001 inj
Drug: Synovian inj — pre-filled syringe
  Arms: Synovian inj

SUMMARY:
This is a randomized, double-blind, multicenter, non-inferiority, pivotal clinical trial to assess the efficacy and safety of the novel hexamethylenediamine (HMDA) cross-linked hyaluronate intra-articular injection (SP5M001) compared with an active comparator, the 1,4-butanediol diglycidyl ether (BDDE) cross-linked hyaluronate (Synovian) in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 40 years or older as of the date of written consent
2. Subject with knee osteoarthritis whose X-ray test results within 6 months from the screening or at the screening visit correspond to grades I - III of the Kellgren & Lawrence scale
3. Subject diagnosed with unilateral or bilateral knee osteoarthritis according to the clinical diagnostic criteria of the American College of Rheumatology (ACR) at screening who have knee joint pain and meet three or more of the following conditions

   * Over 50 years of age

     * Less than 30 minutes of morning stiffness ③ Crepitus on active motion ④ Bony tenderness ⑤ Bony enlargement ⑥ No palpable warmth of synovium
4. Weight bearing pain (WBP) of at least one of both knee joints on 100 mm-VAS ≥ 40 mm when measured at screening and baseline [However, if both sides have symptoms, the knee joint with the higher WBP becomes the joint for evaluation, and the selected joint cannot be changed during the study period.]
5. Walk without relying on a walking aid such as a walker or cane (patients who have been using a walking aid every day since 6 months prior to the screening visit can use the walking aid, and must use the walking aid in the same way throughout the study period.)
6. Ability to fully understand and complete the safety and efficacy measurement questionnaire
7. Voluntary decision for participation and provision of written consent to comply with the precautions after hearing and fully understanding the detailed explanation of the purpose, method, and effects of this study

Exclusion Criteria:

1. Body mass index (BMI) ≥ 35 kg/m2 at screening
2. Hip osteoarthritis or osteoarthritis of another joint that is severe enough to preclude evaluation of knee osteoarthritis at the time of screening
3. Having the following diseases that may affect the efficacy and safety evaluation but not being limited to the following

   * Septic arthritis, rheumatoid arthritis, gout, recurrent pseudogout arthritis, trauma that may damage joint cartilage, congenital abnormalities, calcium deposition disease, diabetes, ochronosis, hemochromatosis, acromegaly, Wilson's disease, primary osteochondrosis, genetic diseases (e.g., hyperkinesis), secondary osteoarthritis caused by collagen gene abnormalities, etc.
   * Sudek's atrophy or severe painful diseases such as Paget's disease
4. Infection or skin disease in the joint area that is unsuitable for injection at the time of screening

   * 5) Active or suspected knee joint infection at the time of screening
   * 6) Complete loss of the Patello-femoral joint space
   * 7) Received the following treatments within 14 days of the screening visit (except those who have passed a 14-day wash-out) or scheduled to be administered during the study period
   * Taking medicines containing ingredients such as glucosamine, chondroitin sulfate, and diacerhein
   * Taking herbal medicines and herbal medicines for osteoarthritis
   * Taking anti-inflammatory painkillers, non-steroidal anti-inflammatory drugs (NSAIDs, prescription/non-prescription drugs), etc. (administration of acetaminophen allowed if passing a 3 day wash-out)
   * Taking oral steroids
   * Hospital physical therapy or oriental medicine treatment (cupping, acupuncture, moxibustion, etc.)

8) Intra-articular injection, such as intra-articular corticosteroid, at the injection site within 6 months from the time of screening 9) Systemic use of steroids within 3 months from the time of screening (including inhalants, however, topical application is permitted only on the upper body) 10) Hyaluronic acid intra-articular injection administered to the injection site within 6 months from the time of screening 11) Surgical operations such as knee joint replacement, including arthroscopic surgery, at the administration site within 6 months from the time of screening; or expecting surgery within 10 months 12) History of artificial joint surgery on the knee joint subject for evaluation 13) Knee joint subject for evaluation diagnosed as Kellgren Lawrence grade 4 within 6 months from the time of screening 14) Moderate or severe joint effusion by Patella tap test at the screening visit 15) History of hypersensitivity to ingredients of the IP or active control drug 16) Antiplatelet agents (excluding aspirin of 300 mg/day or less), heparin, oral anticoagulants (coumarin anticoagulants, thrombin inhibitors, Factor Xa inhibitors, etc.), and thrombolytics must be used during the study 17) Clinically significant abnormalities in liver function (3 times or more than the upper limit of normal for ALT/AST) or abnormalities in renal function (3 times or more than the upper limit of normal for serum creatinine), or severe liver or renal disease at the discretion of the investigator which is judged to have an impact on the effectiveness and safety evaluation of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Change in [Weight-Bearing Pain (WBP)-100mm-visual analogue scale (VAS)] at Week 12 from baseline (visit 2) | week 12
  * Weight Bearing Pain (WBP) - 100mm-visual analogue scale (VAS)

SECONDARY OUTCOMES:
Changes in the following at each visit : Weight Bearing pain(WBP) (Weeks 2, 6, 24, and 36) from baseline (Visit 2) | week 2, 6, 24, 36
  Outcome Measurement of Weight Bearing pain(WBP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Rest pain (RP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Rest pain (RP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Night pain (NP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Night pain (NP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Motion pain (MP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Motion pain (MP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Patient Global Assessment(PGA) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Patient Global Assessment(PGA): 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Investigator Global Assessment (IGA) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Investigator Global Assessment (IGA) : 100mm-visual analogue scale (VAS)
Changes in the following at each visit : Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total score and individual score evaluation (Pain, function, stiffness) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2, 6, 12, 24, 36
  Outcome Measurement of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total score and individual score evaluation (Pain, function, stiffness)
  : WOMAC-Likert Assessment (5-point Likert scale)
Physical assessments at each post-administration visit: Swelling (Weeks 2, 6, 12, 24, and 36) | week 2, 6, 12, 24, 36
  Outcome Measurement of Swelling: 4-point scale
  *4-point scale: 0(none)/1(mild)/2(moderate)/3(severe)
Physical assessments at each post-administration visit: joint-line tenderness on pressure (Weeks 2, 6, 12, 24, and 36) | week 2, 6, 12, 24, 36
  Outcome Measurement of joint-line tenderness: 4-point scale
  *4-point scale: 0(none)/1(mild)/2(moderate)/3(severe)
Physical assessments at each post-administration visit: range of motion (Weeks 2, 6, 12, 24, and 36) | week 2, 6, 12, 24, 36
  The angle was recorded as is for the range of motion.
Proportion of participants who took rescue medication at each post-administration visit and dose of rescue medication (Weeks 2, 6, 12, 24, and 36) | week 2, 6, 12, 24, 36
Post-administration response rate A. Proportion at which WBP decreases by at least 20 mm or improves by at least 40% from baseline at the time of evaluation (B section-Description) | week 2, 6, 12, 24, 36
  *B. Response rate of OMERACT-OARSI (Outcome Measures in Rheumatology-Osteoarthritis Research Society International) I. At least 50% improvement in WOMAC pain or function at the time of evaluation; or at least a 20 point improvement from baseline; or II. meeting 2 of the 3 conditions below
  * At least 20% improvement in WOMAC pain, at least a 10 point improvement from each baseline
  * At least 20% improvement in WOMAC function, at least a 10 point improvement from each baseline
  * At least 20% improvement in patient's global assessment (100 mm-VAS) and at least a 10 point improvement from each baseline

OTHER OUTCOMES:
The incidence rate of Pre-treatment AEs | From week 0 to week 36
The incidence rate of Solicited Local AEs | From week 0 to week 36
The incidence rate of treatment-emergent adverse event (TEAE) | From week 0 to week 36
The incidence rate of Serious TEAEs | From week 0 to week 36
The incidence rate of Serious TEAEs leading to Drug withdrawn | From week 0 to week 36
The incidence rate of Serious TEAEs leading to Death | From week 0 to week 36
The incidence rate of abnormal CS at Post-Treatment on Laboratory | From week 0 to week 36
The incidence rate of abnormal CS at Post-Treatment on Electrocardiogram | From week 0 to week 36
The incidence rate of abnormal on Physical Examination | From week 0 to week 36

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Yeungnam University Medical Center, Daegu
  - Cheonam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Chungnam National University Hospital, Sejong
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Chung-ang University Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyunghee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim KI, In Y, Choi HS, Lee JH, Sim JA, Lee HJ, Moon YW, Shon OJ, Seon JK, Kim YM, Song SJ, Chang CB, Han HS. A Multicentre, Double-Blind, Randomised, Non-Inferiority Trial of a Novel Single-Injection Intra-Articular HMDA-Cross-Linked Hyaluronate Gel for Knee Osteoarthritis. J Clin Med. 2025 Jun 19;14(12):4384. doi: 10.3390/jcm14124384. PMID 40566128